CLINICAL TRIAL: NCT06249958
Title: Transforming Rehabilitation: Personalised Care for a Better Quality of Life (PREPARE, 1st Part)
Brief Title: Transforming Rehabilitation: Personalised Care for a Better Quality of Life
Acronym: PREPARE
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: PREPARE
Record Dates: First submitted 2024-01-09; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis Secondary; Osteoarthritis Primary; Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rehabilitation — Specific rehabilitation exercises
Other: Verticalisation — Day of patient verticalisation after surgery

SUMMARY:
General aim of the project: building and validating an Artificial Intelligence (AI)-based prediction model on rehabilitation outcomes (total joint replacement - TJR - of the hip and knee for primary and secondary osteoarthritis)

Purpose of this specific approval request: identifying data from patients admitted for total joint replacement surgery (hip and knee) at Istituto di Ricerca e Cura a Carattere Scientifico (IRCCS) Istituto Ortopedico Galeazzi (IOG) in 2019 and subsequently discharged to inpatient rehabilitation in the same institution.

DETAILED DESCRIPTION:
The aim is to collect data from patients undergoing elective TJR (baseline, intervention, outcomes) in order to generate and train an AI algorithm.

Patient characteristics (diagnosis, sex, age, American Society of Anesthesiologists (ASA) score, profession, haemoglobin levels, pain, functional autonomy, care giver presence at home), intervention characteristics (surgical procedure, day of surgery, duration of surgery, infection occurrence, need of transfusion, length of hospital stay, verticalization day, rehabilitation program) and outcomes (Barthel Index, functional independence measures, care burden, Patient Reported Outcomes - PROs - when available ) are collected by the Principal Investigator in a dedicated Excel sheet.

The dataset includes information from the entire perioperative care:

* Pre-surgery
* Surgical procedure
* Inpatient rehabilitation
* Post discharge, if available, at 3,6,12,24,60 months.

Such new dataset will by employed to enable a software whose goal is to provide a predictive model for rehabilitation outcomes, which future application would be helping clinicians design evidence-based, personalized rehabilitation programs. The software will be developed by dedicated data science partners within the European Health and Digital Executive Agency (HADEA) research Project n. 101080288, PREPARE.

The study will include elective prosthetic surgery (TJR of the hip and knee) performed in 2019 (January-December) and the subsequent inpatient rehabilitation program.

Data collection will start after approval from the Ethical Committee (EC) and the new dataset must be available before spring 2024. However, retrieving further data may result necessary by general project needs which are currently not entirely foreseeable, therefore we ask authorization for the entire study duration of four years.

Inclusion criteria:

* Patients admitted for inpatient surgery at IOG in 2019 (January-December) and subsequently discharged to inpatient rehabilitation in the same structure.
* Ages ≥18 years
* International Classification of Disease, Ninth Revision, Clinical Modification (ICD-9CM) Diagnoses: 715.15, 16, 25, 26 (primary and secondary osteoarthritis of the hip and knee)
* ICD-9CM Surgical procedures: 81.51, 81.54 (total joint replacement of the hip and knee).

No exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for inpatient surgery at IRCCS Galeazzi Orthopedic Institute in 2019 (January-December) and subsequently discharged to inpatient rehabilitation in the same structure.
* Ages ≥18 years
* International Classification of Disease, Ninth Revision, Clinical Modification (ICD-9CM) Diagnoses: 715.15, 16, 25, 26 (primary and secondary osteoarthritis of the hip and knee)
* ICD-9CM Surgical procedures: 81.51, 81.54 (total joint replacement of the hip and knee).

Exclusion Criteria: N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing a) hip or knee prostethic surgery after primary or secondary osteoarthritis at Galeazzi Orthopedic Hospital, year 2019; b) subsequent inpatient rehabilitation at the same facility.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2027-01-08 (Estimated)

PRIMARY OUTCOMES:
Barthel Index Total score | through study completion, within four years
  0-100, the higher, the better
Functional autonomy measure (total score) | through study completion, within four years
  0-126, the higher, the better
Standard hospital evaluation of patient gait | through study completion, within four years
  Autonomous, autonomous maximum 50 metres, or non autonomous.
Standard hospital evaluation of walking aids needed by the patient | through study completion, within four years
  Crutches, stick, walker.
Standard hospital evaluation of place of discharge | through study completion, within four years
  Home with relatives, home alone, residential care facility.
Standard hospital evaluation of care burden at discharge | through study completion, within four years
  Less than 6 hours a day; less than 3 hours a day; no burden.
Patient-reported outcomes | through study completion, within four years
  Visual Analog Scale (VAS), 0-10, the higher, the better; Short-Form 12, Physical and Mental Scores, 0-100, the higher, the better; Euro QOL - 5 Dimension (EQ-5D), 0-100, the higher, the better; Hip Disability and Osteoarthritis Outcome Score (HOOS), 0-100, the higher, the better; Knee Injury and Osteoarthritis Outcome Score (KOOS), 0-100, the higher, the better.
Functional autonomy measure subdomains | through study completion, within four years
  Mobility, 3-21, the higher, the better; Cognition, 3-21, the higher, the better.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi Sant'Ambrogio, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No